CLINICAL TRIAL: NCT06747936
Title: A Randomized, Double-blind, Active-controlled, Multi-center, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of Combined Administration of AD-2281 and AD-2282 in Patients with Primary Hypercholesterolemia.
Brief Title: A Study to Evaluate the Efficacy and Safety of Co-administration of AD-2281 and AD-2282
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AD-228P3
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AD-2281 + AD-2282 (Experimental)
  Interventions: Drug: AD-2281; Drug: AD-2282
- AD-2281 + Placebo of AD-2282 (Active Comparator)
  Interventions: Drug: AD-2281; Drug: Placebo of AD-2282

INTERVENTIONS:
Drug: AD-2281 — PO, Once daily, 8weeks
Drug: AD-2282 — PO, Once daily, 8weeks
  Arms: AD-2281 + AD-2282
Drug: Placebo of AD-2282 — PO, Once daily, 8weeks
  Arms: AD-2281 + Placebo of AD-2282

SUMMARY:
The purpose of this study is to evaluate the efficacy and safetyof co-administration of AD-2281 and AD-2282 in patients with Primary Hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients with Primary Hypercholesterolemia
* Other inclusions applied

Exclusion Criteria:

* Patients with Secondary Hypercholesterolemia
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change rate of LDL-C | from baseline at 8 weeks
  Percent change (%) of LDL-C from baseline at week 8

IPD SHARING:
Plan to Share IPD: No